CLINICAL TRIAL: NCT03846167
Title: Imaging of Primary or Recurrent Breast Cancer With 18F-FluorThanatrace Positron Emission Tomography (PET/CT)
Brief Title: Imaging of Primary or Recurrent Breast Cancer With 18F-FluorThanatrace PET/CT
Acronym: FTT 2
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 832165
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue will only be collected for research purpose, if there is adequate tissue available, after the clinical diagnostic needs are met.
  If the participants are undergoing a clinical biopsy for suspected breast cancer, they may be asked to provide additional samples for experimental pathologic evaluations or establishment of cell lines at the time of the clinical biopsy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FTT PET/CT: The imaging procedure may include one or both of the following imaging sessions; 1) a 45- 60 minute dynamic scan, starting at approximately the same time as the injection and/or 2) a skull base to mid-thigh scan starting approximately 60 minutes post injection of [18F]FTT.
  Participants will be asked to complete the following research procedures: [18F]FTT PET/CT scan before surgery or treatment [18F]FTT PET/CT scan after you start treatment (optional)
  Interventions: Drug: Imaging Drug FluorThanatrace (FTT)

INTERVENTIONS:
Drug: Imaging Drug FluorThanatrace (FTT) — [18F]FTT is an investigational radioactive PET drug used to see PARP-1 activity in tumors. This radioactive imaging drug is injected into the body to see how it goes into places where there is active breast cancer. Using an imaging scan called Positron Emission Tomography (PET/CT), the radioactive drug can be seen in the body.

SUMMARY:
Patients with known or suspected, in the opinion of an investigator, primary or metastatic breast cancer may be eligible for this study. Up to 45 evaluable participants may undergo study imaging in this protocol. The imaging procedure may include one or both of the following imaging sessions; 1) a 45- 60 minute dynamic scan, starting at approximately the same time as the injection and/or 2) a skull base to mid-thigh scan starting approximately 60 minutes post injection of [18F]FTT. The planned scanning protocol will be selected by an investigator and will be discussed with the participant prior to the imaging visit. The PET/CT scan will include an injection of [18F]FTT. Data will be collected to evaluate uptake of [18F]FTT in breast cancer and compare with PARP-1 activity in tissue, when available. If participants are getting neoadjuvant or other systemic therapy, a second optional scan may be performed 1 day to 4 weeks after therapy begins to evaluate whether response correlates with increase in PARP-1 activity.

DETAILED DESCRIPTION:
Patients who come to the clinical practices of the University of Pennsylvania for diagnosis and/or treatment of a known or suspected breast cancer and who meet the study inclusion criteria may be approached by study staff for recruitment into this study. Eligibility criteria will be checked and study personnel will provide a copy of the approved consent form to the potential subject. Patients will be approached initially in person, by phone or email about study participation. The patient will be given an opportunity to go over the consent form and have any questions answered by study staff or a study investigator. After discussion of the study procedures, risks and benefits, if the patient agrees to participate in the study, the [18F]FTT PET/CT will be ordered by a physician and scheduled. Patients may cancel the scan appointment at any time prior to the injection of [18F]FTT with no negative impact to them or their medical care at UPenn. A written informed consent will be reviewed with the patient and signed prior to any study procedures being performed. Participants may withdraw from the study at any time at their own request, or they may be withdrawn at any time at the discretion of the investigator or sponsor for safety, behavioral, or administrative reasons. If a participant does not return for a scheduled visit, every effort will be made to contact the subject.

Women of childbearing potential will have a urine pregnancy test performed within 1 day prior to injection of [18F]FTT.

The baseline [18F]FTT PET/CT will take place prior to surgical resection of a primary breast cancer, or before starting therapy. Adverse event follow up after the PET/CT scan may occur by telephone or in person, depending on the participant's schedule. Follow up will take place the next available business day (i.e. not a weekend or a holiday). The adverse event monitoring period is 24 hours following [18F]FTT injection.

An optional post-therapy [18F]FTT PET/CT may occur approximately 1 day to 4 weeks after the start of new therapy regimen.

Participants will be asked to give consent to allow for collection of pathology tissue for use in this research study. Archival tissue may be collected from an existing tissue sample. Additional tissue may be collected during a clinical biopsy or surgical procedure, if a procedure is scheduled as part of their clinical care or, it can be collected for research purposes only, if the patient has consented for this additional collection.

Participants will be asked permission to access their medical records for follow up of their clinical care and treatment as part of the consent for this study.

Long term follow up will occur by medical record review for the duration of the participant's cancer care until death or 15 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 18 years of age
2. Known or suspected, in the opinion of an investigator, primary breast or metastatic breast cancer. For subjects with primary breast cancer we will target lesion size of 1.0 cm or greater on at least one type of standard imaging.
3. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who are pregnant or breast feeding at the time of enrollment will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential prior to FTT injection.
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
3. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who come to the clinical practices of the University of Pennsylvania for diagnosis and/or treatment of a known or suspected breast cancer and who meet the study inclusion criteria may be approached by study staff for recruitment into this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
PARP-1 Activity in Breast Cancer | 4 Years
  Evaluate PARP-1 activity in breast cancer using measures of uptake of [18F]FluorThanatrace.

SECONDARY OUTCOMES:
Activity in Tissues | 4 Years
  Correlate [18F]FluorThanatrace uptake measures with PARP-1 pathology assays of activity in tissue.
Hormone Receptor Status | 4 Years
  Correlate [18F]FluorThanatrace uptake measures with hormone receptor status.
Change After Therapy | 4 Years
  Determine whether [18F]FluorThanatrace uptake measures change after therapy start.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonald ES, Pantel AR, Shah PD, Farwell MD, Clark AS, Doot RK, Pryma DA, Carlin SD. In vivo visualization of PARP inhibitor pharmacodynamics. JCI Insight. 2021 Apr 22;6(8):e146592. doi: 10.1172/jci.insight.146592. PMID 33884961